CLINICAL TRIAL: NCT01168986
Title: The Effectiveness of a Mechanical Manual Therapy Device in the Treatment of Neck Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 340-2009; 340-2009 (Other: University of Florida)
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-05

CONDITIONS: Neck Pain
Keywords: neck pain; manual therapy; exercise
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pulstar Multiple Impulse Therapy (Active Comparator): Use of the PulStar Multiple Impulse Therapy (Sense Technology). A mechanical manual therapy device.
  Interventions: Other: Pulstar Multiple Impulse Therapy
- Exercise (Active Comparator): Participants perform an exercise to strengthen the deep neck flexors
  Interventions: Other: Exercise
- No intervention (No Intervention): Participants receive/perform no intervention

INTERVENTIONS:
Other: Pulstar Multiple Impulse Therapy — Use of the PulStar Multiple Impulse Therapy (Sense Technology). A mechanical manual therapy device.
  Arms: Pulstar Multiple Impulse Therapy
Other: Exercise — Participants perform an exercise to strengthen the deep neck flexors
  Arms: Exercise

SUMMARY:
This study is comparing the effectiveness of a mechanical manual therapy device to a specific exercise to no treatment in individuals experiencing neck pain. We are interested in the effects of the interventions on neck pain, disability related to neck pain, and pain sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* currently experiencing neck pain which does not extend below the elbow
* pain at least 4/10 over the past 24 hours
* appropriate for conservative management of neck pain
* english speaking

Exclusion Criteria:

* surgery to the neck within the past 6 months
* systemic problem know to affect sensation
* other chronic pain condition other than neck pain
* neck pain as the result of trauma such as whiplash
* neck pain as the result of a fracture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2009-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel E Bialosky, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulstar Multiple Impulse Therapy | Exercise | No Intervention
Started | 20 | 21 | 21
Completed | 18 | 20 | 21
Not Completed | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulstar Multiple Impulse Therapy | Exercise | No Intervention | Total
Number analyzed (Participants) | 20 | 21 | 21 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.15 (12.32) | 31.48 (10.95) | 36.33 (14.12) | 33.98 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 16 | 47
  Male | 4 | 6 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 18 | 19 | 19 | 56
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 4 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 4 | 8
  White | 11 | 15 | 15 | 41
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 21 | 62

OUTCOME MEASURES:

1. Primary Outcome: 2 Week Change in Pain Score on a Numeric Rating Scale
Description: a 101 point numeric rating scale of neck pain with 0 indicating no pain at all and 100 indicating the worst pain imaginable
Time Frame: 2 weeks
Population: The numbers of participants analyzed is not consistent with number of participants enrolled in the study due to missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulstar Multiple Impulse Therapy | Exercise | No Intervention
Number analyzed (Participants) | 18 | 19 | 19
units on a scale | 6.39 (24.23) | 20.37 (23.67) | 6.45 (19.88)
Statistical Analysis 1: Comparison: Pulstar Multiple Impulse Therapy vs Exercise vs No Intervention; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis

2. Primary Outcome: 2 Week Change in Disability on the Neck Disability Index
Description: A functional questionnaire (the neck disability index) to assess self report of disability related to neck pain. The neck disability index is a 10 item questionnaire assessing neck pain related disability. Items are scored from 0 to 5 with the total score doubled resulting in a final score from 0 to 100 with higher scores indicating higher levels of perceived disability.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 2 week change in units a scale
Arm/Group | Pulstar Multiple Impulse Therapy | Exercise | No Intervention
Number analyzed (Participants) | 18 | 20 | 19
2 week change in units a scale | 4.44 (8.53) | 5.50 (9.53) | 0.42 (8.37)
Statistical Analysis 1: Comparison: Pulstar Multiple Impulse Therapy vs Exercise vs No Intervention; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis

3. Primary Outcome: Immediate Change in Pain Sensitivity Using a Numeric Pain Rating Scale
Description: Participants rated the pain associated with a standardized (51 degrees Celsius) thermal stimulus applied to the plantar surface of their dominant foot using a 0 to 100 numeric pain rating scale with 0 indicating no pain at all and 100 indicating the most intense pain sensation imaginable.
Time Frame: Immediate within session change pre to post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulstar Multiple Impulse Therapy | Exercise | No Intervention
Number analyzed (Participants) | 17 | 19 | 18
units on a scale | 0.58 (15.39) | -0.76 (16.66) | 1.62 (10.83)
Statistical Analysis 1: Comparison: Pulstar Multiple Impulse Therapy vs Exercise vs No Intervention; Test type: Superiority or Other; p = 0.87, Mixed Models Analysis

4. Secondary Outcome: Change From Baseline in Neck Extension Range of Motion at 2 Weeks
Description: change in neck extension range of motion over a 2 week period
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pulstar Multiple Impulse Therapy | Exercise | No Intervention
Number analyzed (Participants) | 18 | 19 | 19
degrees | 2.50 (15.46) | 1.32 (9.04) | -1.84 (6.06)
Statistical Analysis 1: Comparison: Pulstar Multiple Impulse Therapy vs Exercise vs No Intervention; Test type: Superiority or Other; p = 0.45, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Pulstar Multiple Impulse Therapy | Exercise | No Intervention
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21

LIMITATIONS AND CAVEATS:
Participants were individuals with neck pain responding to a study and not necessarily seeking care. As a result, the findings may not directly translate to individuals with neck pain seeking care from a healthcare provider.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No